CLINICAL TRIAL: NCT00674271
Title: Immune Profile and Complications Risk in Type 2 Diabetes
Brief Title: Immune Profile and Complication Risk in Type 2 Diabetes
Acronym: IMPACT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20080059
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Mannose-Binding lectin; Toll-Like Receptors; Atherosclerosis; Carotid Arteries; Diabetes Complications; Diabetic Angiopathies
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis; Diabetes Complications; Diabetic Angiopathies

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Whole blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetics: 100 patients with newly diagnosed (<5 years since diagnosis) type 2 diabetes referred from general practitioners to Medical Department M, Aarhus University Hospital, Denmark.
- Controls: 100 healthy (no diabetes or prediabetes in oral glucose tolerance test) control subjects matched for age and gender

SUMMARY:
The aim of this study is to investigate the relation between individual differences in pattern recognition molecules (PRM's) in the innate immune system and the prevalence and development of vascular complications in patients with type 2 diabetes.

This is based on the hypothesis that pattern recognition molecules (PRM's) in the innate immune system contributes to a chronic low grade inflammation in diabetic patients. Variation in PRM's - at the genome, proteome as well as the functional level - are therefore associated with the degree of chronic low grade inflammation, and probably also with the prevalence of vascular complications.

DETAILED DESCRIPTION:
Aim: The primary aims of the project are:

1. By use of advanced magnetic resonance imaging to characterize the prevalence of atherosclerosis in the carotid arteries in patients with newly diagnosed type 2 diabetes.
2. To investigate if individual differences in the innate immune system contributes to the prevalence and development of cardiovascular disease in patients with type 2 diabetes.
3. To prospectively observe the cardiovascular morbidity and mortality in a cohort of patients with type 2 diabetes seen in the light of the obtained baseline characteristics.

Background: Type 2 diabetes is a very common disease in the western world. Patients with type 2 diabetes are at risk of a number of complications, including macroangiopathy which involves an accelerated atherosclerosis, that causes most of the increased mortality and morbidity in type 2 diabetics. Mounting evidence suggests that development of vascular complications is associated to a chronic low grad inflammation in type 2 diabetes. Individual differences in the innate immune system might contribute to this chronic low grade inflammation as it has become apparent that in some situations - as after tissue ischemia or in diabetes - a change in the body's own cell glycosylations occurs, which leads to increased affinity of PRM's. This study will focus primarily on two families of PRM's: Collectins and Toll-like receptors.

Methods: The study consists of a prospective observational cohort study of 100 newly diagnosed type 2 diabetic patients with continuous 2-year clinical follow-up and a register-based follow-up of morbidity and mortality study after 5 and 10 years. Furthermore 100 healthy control subjects will be included. Baseline data will represent a independent cross-sectional study of the relationship between the innate immune system, glycemic control and the presence of atherosclerosis in the carotid arteries in newly diagnosed type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diabetics: Newly diagnosed (<5 years since diagnoses) type 2 diabetes due to national diagnosis criteria
* Controls: No diabetes or prediabetes in oral glucose tolerance test

Both:

* Age > 18 years
* Signed informed consent

Exclusion Criteria:

Both:

* Pacemaker or other magnetic materials in the body
* Severe claustrophobia
* Pregnancy/lactation
* Cancer - former or current
* Acute or chronic infection
* Dialysis-dependent kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients with newly diagnosed (<5 years since diagnosis) type 2 diabetes referred from general practitioners to Medical Department M, Aarhus University Hospital, Denmark.
  100 healthy (no diabetes or prediabetes in oral glucose tolerance test) control subjects matched for age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Plaque burden in carotid arteries | Individual

SECONDARY OUTCOMES:
Serum levels of pattern recognition molecules | Individual
Genotyping genes for pattern recognition molecules | Individual

CONTACTS AND LOCATIONS:
Overall Officials: Jens S Christiansen, Prof., MD, Principal Investigator — Medical Department M, Aarhus University Hospital, Denmark
Locations (1):
- Medical Department M, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Laugesen E, Hoyem P, Fleischer J, Kumarathas I, Knudsen ST, Hansen KW, Christiansen JS, Hansen TK, Poulsen PL. Reduced Subendocardial Viability Ratio Is Associated With Unfavorable Cardiovascular Risk Profile in Women With Short Duration of Type 2 Diabetes. Am J Hypertens. 2016 Oct;29(10):1165-72. doi: 10.1093/ajh/hpw066. Epub 2016 Jul 12. PMID 27405963
- [Derived] Funck KL, Laugesen E, Hoyem P, Fleischer J, Cichosz SL, Christiansen JS, Hansen TK, Poulsen PL. Low Physical Activity Is Associated With Increased Arterial Stiffness in Patients Recently Diagnosed With Type 2 Diabetes. Am J Hypertens. 2016 Jul;29(7):882-8. doi: 10.1093/ajh/hpv197. Epub 2015 Dec 28. PMID 26714500
- [Derived] Fleischer J, Lebech Cichosz S, Hoeyem P, Laugesen E, Loegstrup Poulsen P, Sandahl Christiansen J, Tarnow L, Hansen TK. Glycemic variability is associated with reduced cardiac autonomic modulation in women with type 2 diabetes. Diabetes Care. 2015 Apr;38(4):682-8. doi: 10.2337/dc14-0654. Epub 2015 Jan 8. PMID 25573884
- [Derived] Laugesen E, Hoyem P, Christiansen JS, Knudsen ST, Hansen KW, Argraves WS, Hansen TK, Poulsen PL, Rasmussen LM. Plasma levels of the arterial wall protein fibulin-1 are associated with carotid-femoral pulse wave velocity: a cross-sectional study. Cardiovasc Diabetol. 2013 Jul 18;12:107. doi: 10.1186/1475-2840-12-107. PMID 23866070
- [Derived] Laugesen E, Hoyem P, Stausbol-Gron B, Mikkelsen A, Thrysoe S, Erlandsen M, Christiansen JS, Knudsen ST, Hansen KW, Kim WY, Hansen TK, Poulsen PL. Carotid-femoral pulse wave velocity is associated with cerebral white matter lesions in type 2 diabetes. Diabetes Care. 2013 Mar;36(3):722-8. doi: 10.2337/dc12-0942. Epub 2012 Nov 5. PMID 23129135